CLINICAL TRIAL: NCT06196424
Title: Observational, Prospective, Multicentre Study to Investigate the Family History of Cancer in Patients With Non-small Cell Lung Cancer (FAHIC - Lung).
Brief Title: A Study to Investigate the Family History of Cancer in Patients With Non-small Cell Lung Cancer (FAHIC - Lung).
Acronym: FAHIC-Lung
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Collaborators: A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: 27.23 CET 2 CBM
Record Dates: First submitted 2023-12-19; First posted 2024-01-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: family history of cancer; inherited risk; risk factors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: study questionnaire to investigate family history — Participants will be given a specific study questionnaire (paper-based) to fill at home, which was specifically designed to collect family history information

SUMMARY:
Germline testing to find genetic alteration that can be linked to inherited susceptibility of developing the disease is recommended for patients diagnosed with certain solid cancers, such as breast, prostate and ovarian, due to strong association with inheritable mutations implying familiar counselling. Non-Small Cell Lung Cancer (NSCLC) is the leading cancer-related cause of death and smoking habitude is the main modifiable risk, while environmental factors, such as radon, asbestosis and fine polluting particles account for most diagnoses among never or light smokers. At the same time, the relative risk (RR) of lung cancer correlates with the number of relatives diagnosed with lung cancer.

A recent study of 7788 patients with NSCLC who receiving a germline testing described a prevalence of genetic alterations linked to inherited susceptibility of cancer in 14.9% of cases, highlighting the potential role of genetic However, all the available studies investigating the family history of cancer among patients with NSCLC are retrospective and do not consider modifiable risk factors such as smoking, working habits and geographical origins.

The objective of this study is the detailed description of the family history of cancer among patients with NSCLC and the description of distribution of other risk factors, such as smoking, among the study participants, in order to establish whether there are specific family history clusters that can help clinicians in directing patients to genetic counselling.

The study will enrol consecutive patients with NSCLC, independently from age, disease stage, smoking status, and clinic-pathological characteristics.

Participants will provide clinical anamnestic information filling an ad hoc self-reported study questionnaire, internally validated by the genetic expert of the steering committee. Data of interest include: Family history of cancer; Type of tumours/primary tumour site among relatives with history of cancer; Age at diagnosis among relatives with history of cancer; Biological sex of relatives with history of cancer; Exposure to tobacco smoking and smoking habits among relatives with history of cancer; Geographical origin of participants and relatives with history of cancer; Personal history of multiple malignancies; Potential professional and environmental exposure to carcinogens of participants and relatives with history of cancer; Ethnicity of both participants and relatives with history of cancer.

The study does not require any additional hospital access from the patients since the questionnaire will be returned at the following planned clinical consultation to minimize recall bias.

The investigators will collect the following clinic-pathologic characteristics: Smoking status (active/passive, package/year, total years of smoking); Eastern Cooperative Oncology Group Performance Status (ECOG-PS); Age at diagnosis; Tumour histology; Tumour stage at diagnosis according to the 8th edition of TNM staging system; Ethnicity; Professional and environmental exposure to carcinogens; Programmed death ligand-1 tumour proportion score (PD - L1 TPS); Any available oncogenic drivers including epidermal growth factor receptor (EGFR), Kirsten rat sarcoma virus (KRAS), BRAF, c-MET, mutations and Anaplastic lymphoma kinase (ALK), ROS-1, RET, neurotrophic tyrosine receptor kinase NTRK translocation/gene fusions; Personal history of other synchronous/metachronous primary malignancies.

DETAILED DESCRIPTION:
This is a prospective, observational, multi-centre study. Our study population will be represented by consecutive patients with histologically diagnosed NSCLC, regardless of their age, TNM stage, smoking status, and other clinic-pathologic characteristics.

The primary objectives of this study will be:

* description of the FHC and potential within-family clusters of other risk factors among patients with NSCLC
* identification of potential FHC patterns and within-family clusters of other risk factors to address patient with NSCLC to systematic genetic counselling.

Secondary objectives include:

- description of clinic-pathological and oncological characteristics of patients with NSCLC of according to FHC patterns and within-family clusters of other risk factors.

Participants' history will be carefully collected by investigators through a dedicated self-reported study questionnaire, which has been developed for the purpose of this study (provided as Appendix 1) The ad-hoc study questionnaire has been validated by the genetic expert of the steering committee who will train each investigator to translate the returned questionnaire into standardized family trees.

Study questionnaire will focus on:

* Family history of cancer;
* Type of tumours/primary tumour site among relatives with history of cancer;
* Age at diagnosis among relatives with history of cancer;
* Biological sex of relatives with history of cancer;
* Exposure to tobacco smoking and smoking habits among relatives with history of cancer;
* Geographical origin of participants and relatives with history of cancer;
* Personal history of multiple malignancies;
* Potential professional and environmental exposure to carcinogens of participants and relatives with history of cancer;
* Ethnicity of both participants and relatives with history of cancer.

To minimize risks of recalling bias, patients will be followed up for 4 weeks through 2 study visits: the first study visit at enrolment and the follow-up study visit.

During the first study visit all patient's clinic-pathologic will be collected and study participants will be given the ad-hoc questionnaire, which will be returned to the study personnel at the follow-up study visit.

The following clinic-pathologic characteristics will be collected:

* Smoking status (active/passive, package/year, total years of smoking)
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS)
* Age at diagnosis;
* Tumour histology;
* Tumour stage at diagnosis according to the 8th edition of TNM staging system;
* Ethnicity;
* Professional and environmental exposure to carcinogens;
* Programmed death ligand-1 tumour proportion score (PD - L1 TPS)
* Any available oncogenic drivers including epidermal growth factor receptor (EGFR), Kirsten rat sarcoma virus (KRAS), BRAF, c-MET, mutations and Anaplastic lymphoma kinase (ALK), ROS-1, RET, neurotrophic tyrosine receptor kinase NTRK translocation/gene fusions.

Personal history of other synchronous/metachronous primary malignancies.

Study data will be collected through dedicated electronic case report form (e-CRF). A full list of information that will be collected through the dedicated eCRF (provided as appendix 2).

Even though no established FHC criteria exists to refer patients with NSCLC to a genetic counselling for germ-line testing, investigators will assess participant questionnaire at the follow-up study visit and refer patients to genetic counselling when clinically indicated as per local routine practice.

Following collection of participants' questionnaires, the investigators will be able to reconstruct patients' family three with additional information on how other potential risk factors, such as history of smoking, exposure to professional/environmental carcinogens, segregate within the relatives with history of cancer.

The investigators will be able to describe whether recurrent family clusters of malignancies/risk factors are specifically associated with risk of lung cancer in order to individuate patients to specifically address to systematic genetic counselling, to assess eligibility for germ-line testing in clinical practice. Secondly, the investigators will also assess the distribution of participants clinic-pathologic characteristics to assess whether any patients and/or tumour-related feature is associated with patterns of FHC and within-family clustering of other risk factors.

The esteemed study duration is 24 months. Enrolment will start after protocol approval and will last for 12 months. Data analysis will last 12 months from the closure of data collection.

Statistical Plan and Sample Size

Given the descriptive nature of the study, and the lack of available data on the relationship between family history of cancer and NSCLC, the minimum sample size for the study has been established on the only study available to date which investigated distribution of FHC among unselected patients with stage IV NSCLC, which described a high familiar burden of cancer (i.e. especially enriched FHC with cases of cancer in both the collateral and lineal family lines) in up to the 6.8% of patients [14]. On the basis of this data, the investigators hypothesized a prevalence of 10% of participants with an especially enriched family history of cancer in our study population; assuming a confidence level of 95% with a total width for the confidence interval of 0.1 (precision of +/- 5%) and considering a 10% drop out, the minimum number of subjects that will need to be enrolled to properly describe the group of interest following a binomial "exact" calculation of the sample size is 175 Descriptive statistics will be used as appropriate to report FHC data, distribution of within-family other risk factors and baseline clinic-pathologic characteristics. The Fisher exact test and the χ2 test will be used as appropriate to compare categorical variables (e.g. distribution of baseline characteristics according to the personal/familial positive or negative history). Analyses were performed using the R-studio software, R Core Team (2021). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria, and the MedCalc® Statistical Software version 20 (MedCalc Software Ltd, Ostend, Belgium; https://www.medcalc.org; 2021).

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of Non-Small Cell Lung Cancer (all stages)
* Age ≥ 18 years old
* Signed informed consent
* Availability of familiar and/or personal anamnestic data of cancer

Exclusion Criteria:

* Unavailability of familiar and/or personal anamnestic data of cancer
* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, observational, multi-centre study. Our study population will be represented by consecutive patients with histologically diagnosed NSCLC, regardless of their age, TNM stage, smoking status, and other clinic-pathologic characteristics.
  Patients' history will be carefully collected by investigators through a dedicated self-reported study questionnaire, which has been developed for the purpose of this study (provided as Appendix 1).
  The ad-hoc study questionnaire has been validated by the genetic expert of the steering committee who will train each investigator to translate the returned questionnaire into standardized family trees.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
family history of cancer among participants | through study completion, an average of 1 year
  The study questionnaire will collect information on: family history of cancer, type of primary tumors among relatives and age at diagnosis, biological sex, exposure to tobacco smoking, geographical origin, potential professional and environmental exposure, ethnicity

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
  - AOU Citta della Salute le Molinette, Torino

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared and there is no plan at this stage. Future requests will be considered upon reasonable requests. Fully anonymised data will be considered for sharing after assessment of the study PI, data protection office of the sponsor and with a data trasnfer agreement in place.

REFERENCES:
- [Result] Stjepanovic N, Moreira L, Carneiro F, Balaguer F, Cervantes A, Balmana J, Martinelli E; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Hereditary gastrointestinal cancers: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-updagger. Ann Oncol. 2019 Oct 1;30(10):1558-1571. doi: 10.1093/annonc/mdz233. No abstract available. PMID 31378807
- [Result] Malvezzi M, Santucci C, Boffetta P, Collatuzzo G, Levi F, La Vecchia C, Negri E. European cancer mortality predictions for the year 2023 with focus on lung cancer. Ann Oncol. 2023 Apr;34(4):410-419. doi: 10.1016/j.annonc.2023.01.010. Epub 2023 Mar 6. PMID 36882139
- [Result] Steuer CE, Jegede OA, Dahlberg SE, Wakelee HA, Keller SM, Tester WJ, Gandara DR, Graziano SL, Adjei AA, Butts CA, Ramalingam SS, Schiller JH; ECOG-ACRIN 1505 Investigators. Smoking Behavior in Patients With Early-Stage NSCLC: A Report From ECOG-ACRIN 1505 Trial. J Thorac Oncol. 2021 Jun;16(6):960-967. doi: 10.1016/j.jtho.2020.12.017. Epub 2021 Feb 1. PMID 33539971
- [Result] Malhotra J, Malvezzi M, Negri E, La Vecchia C, Boffetta P. Risk factors for lung cancer worldwide. Eur Respir J. 2016 Sep;48(3):889-902. doi: 10.1183/13993003.00359-2016. Epub 2016 May 12. PMID 27174888
- [Result] Riudavets M, Garcia de Herreros M, Besse B, Mezquita L. Radon and Lung Cancer: Current Trends and Future Perspectives. Cancers (Basel). 2022 Jun 27;14(13):3142. doi: 10.3390/cancers14133142. PMID 35804914
- [Result] Cannon-Albright LA, Carr SR, Akerley W. Population-Based Relative Risks for Lung Cancer Based on Complete Family History of Lung Cancer. J Thorac Oncol. 2019 Jul;14(7):1184-1191. doi: 10.1016/j.jtho.2019.04.019. Epub 2019 May 7. PMID 31075544
- [Result] Ji J, Sundquist J, Sundquist K, Zheng G. Familial risk associated with lung cancer as a second primary malignancy in first-degree relatives. BMC Cancer. 2022 Oct 12;22(1):1057. doi: 10.1186/s12885-022-10149-7. PMID 36224547
- [Result] Chang ET, Smedby KE, Hjalgrim H, Glimelius B, Adami HO. Reliability of self-reported family history of cancer in a large case-control study of lymphoma. J Natl Cancer Inst. 2006 Jan 4;98(1):61-8. doi: 10.1093/jnci/djj005. PMID 16391372
- [Result] Murff HJ, Spigel DR, Syngal S. Does this patient have a family history of cancer? An evidence-based analysis of the accuracy of family cancer history. JAMA. 2004 Sep 22;292(12):1480-9. doi: 10.1001/jama.292.12.1480. PMID 15383520
- [Result] Cortellini A, Giusti R, Filetti M, Citarella F, Adamo V, Santini D, Buti S, Nigro O, Cantini L, Di Maio M, Aerts JGJV, Bria E, Bertolini F, Ferrara MG, Ghidini M, Grossi F, Guida A, Berardi R, Morabito A, Genova C, Mazzoni F, Antonuzzo L, Gelibter A, Marchetti P, Chiari R, Macerelli M, Rastelli F, Della Gravara L, Gori S, Tuzi A, De Tursi M, Di Marino P, Mansueto G, Pecci F, Zoratto F, Ricciardi S, Migliorino MR, Passiglia F, Metro G, Spinelli GP, Banna GL, Friedlaender A, Addeo A, Ficorella C, Porzio G, Tiseo M, Russano M, Russo A, Pinato DJ. High familial burden of cancer correlates with improved outcome from immunotherapy in patients with NSCLC independent of somatic DNA damage response gene status. J Hematol Oncol. 2022 Jan 21;15(1):9. doi: 10.1186/s13045-022-01226-2. PMID 35062993
- [Result] Benusiglio PR, Fallet V, Sanchis-Borja M, Coulet F, Cadranel J. Lung cancer is also a hereditary disease. Eur Respir Rev. 2021 Oct 20;30(162):210045. doi: 10.1183/16000617.0045-2021. Print 2021 Dec 31. PMID 34670806
- [Result] Sorscher S, LoPiccolo J, Heald B, Chen E, Bristow SL, Michalski ST, Nielsen SM, Lacoste A, Keyder E, Lee H, Nussbaum RL, Martins R, Esplin ED. Rate of Pathogenic Germline Variants in Patients With Lung Cancer. JCO Precis Oncol. 2023 Sep;7:e2300190. doi: 10.1200/PO.23.00190. PMID 37992258

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT06196424/Prot_SAP_000.pdf